CLINICAL TRIAL: NCT01545193
Title: The Effect of Age on the Incidence of Postoperative Residual Neuromuscular Blockade
Status: Completed | Type: Observational
Sponsor: Endeavor Health (Other)
Responsible Party: Principal Investigator, Glenn Murphy, Director, Cardiac Anesthesia and Clinical Research, Endeavor Health
Other Study IDs: EH11-045
Record Dates: First submitted 2012-03-01; First posted 2012-03-06 (Estimated); Results first posted 2015-04-06 (Estimated); Last update posted 2019-09-16 (Actual); Status verified 2019-09

CONDITIONS: Residual Neuromuscular Blockade in Elderly Patients
Keywords: Elderly; Residual neuromuscular blockade
MeSH Terms: conditions — Delayed Emergence from Anesthesia | interventions — Aging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Age 18-50: This is a younger study cohort who is anticipated to have a lower incidence of residual neuromuscular blockade
  Interventions: Other: Age and incidence of residual neuromuscular blockade
- Age 70-90: This is a older study cohort who is anticipated to have a higher incidence of residual neuromuscular blockade
  Interventions: Other: Age and incidence of residual neuromuscular blockade

INTERVENTIONS:
Other: Age and incidence of residual neuromuscular blockade — An older cohort is anticipated to have a higher incidence of residual neuromuscular blockade

SUMMARY:
Residual neuromuscular blockade is frequently observed in the early postoperative period when patients have received a general anesthetic with muscle relaxants. At the present time it is uncertain whether certain patient populations are at greater risk for this common anesthetic complication. However, it is possible that elderly surgical patients may exhibit a higher incidence of residual neuromuscular blockade. The aim of this clinical trial is to determine the incidence of residual neuromuscular blockade in a cohort of younger (ages 18-50) and older (ages 70-90) patients undergoing surgery and general anesthesia.

DETAILED DESCRIPTION:
300 patients will be enrolled in this study. Patients will be selected for enrollment by reviewing the operating room schedule on the day prior to the procedure. Two groups of patients will be examined; group 1 will consist of patients ages 18-50 (n=150) and group 2 will consist of patients age 70-90 (n=150). Patients will be enrolled in blocks of 20 to ensure an equal distribution of subjects in each age group over time.

Anesthetic and neuromuscular management will be standardized in both study cohorts

Neuromuscular Monitoring:

On arrival to the PACU, a blinded research assistant will obtain a quantitative TOF measurement in all subjects. The TOF-Watch SX will be used to obtain these measurements. Two consecutive responses to TOF stimulation (separated by > 15 seconds) will be obtained, and the average of the two values recorded. If the measurements differ by greater than 10%, additional TOF ratios can be obtained (up to a total of 4 TOF values), and the closest two ratios averaged. The number of patients with TOF ratios < 0.7, 0.8, and 0.9 (which are levels of residual neuromuscular block associated with various adverse clinical outcomes) in each group will be compared.

Signs and Symptoms of Residual Neuromuscular Blockade After TOF data is collected on arrival to the PACU, the patients will be carefully examined for signs and symptoms of muscle weakness by a blinded research assistant. A standardized examination form will be used to determine the presence or absence of muscle weakness in a variety of muscle groups. The examination will be performed on arrival to the PACU and again 15 minutes after admission.

Respiratory Events Potentially Related to Residual Neuromuscular Blockade

Pulse oximetry will be used to continuously monitor arterial oxygen saturations (Sp02) during patient transport and in the PACU. Patients will be transported to the PACU without supplemental oxygen (unless the anesthesia care provider determines that oxygen therapy is required for patient safety-per standard practice). All patients will be placed on 2 liters nasal cannula oxygen in the PACU. In the PACU, pulse oximetry will be used to continuously measure Sp02. Oxygenation data will be stored and recorded every minute for the first 30 minutes of the PACU admission. In addition to oxygenation data, patients will be assessed during transportation to the PACU and during the first 30 minutes of the PACU admission for evidence of airway obstruction.

PACU Length of Stay The impact of age and residual blockade on length of PACU stay will be determined. The time required to meet discharge criteria and achieve actual discharge will be noted.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting for elective surgical procedures with an expected duration greater than 45 minutes.
* ASA I to III patients ≥ 18 years of age, presenting for surgery requiring maintenance of neuromuscular blockade in the operating room, will be eligible for enrollment.

Exclusion Criteria:

1. presence of an underlying neuromuscular disease
2. use of drugs known to interfere with neuromuscular transmission (antiseizure medications, anticholinesterases, magnesium sulfate)
3. renal insufficiency (serum creatinine > 1.8 mg/dL) or renal failure.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing general anesthesia and surgery
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2011-06; Primary Completion 2013-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Glenn S. Murphy, MD, Principal Investigator — Endeavor Health
Locations (1):
- NorthShore University HealthSystem, Evanston, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Age 18-50 | Age 70-90
Started | 150 | 150
Completed | 150 | 149
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Age 18-50 | Age 70-90 | Total
Number analyzed (Participants) | 150 | 149 | 299
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 150 | 0 | 150
  >=65 years | 0 | 149 | 149
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 38 [30 to 46] | 75 [72 to 80] | 57 [51 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 98 | 84 | 182
  Male | 52 | 65 | 117
Region of Enrollment [Number; unit: participants]
  United States | 150 | 149 | 299

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Residual Neuromuscular Blockade
Description: The TOF-Watch SX will be used to determine the incidence of residual neuromuscular blockade. The TOF-Watch SX consists of a nerve stimulator and a sensor to quantify the TOF ratio. Two consecutive responses to train-of-four (TOF) stimulation will be obtained, and the average of the two values recorded. If the measurements differ by greater than 10%, additional TOF ratios can be obtained (up to a total of 4 TOF values), and the closest two ratios averaged. The number of patients with TOF ratios < 0.9 in each group will be compared.
Time Frame: Early postoperative period, up to 24 hours
Measure: Number; unit: participants
Arm/Group | Age 18-50 | Age 70-90
Number analyzed (Participants) | 150 | 149
participants | 45 | 86

2. Secondary Outcome: Signs and Symptoms of Residual Neuromuscular Blockade
Description: A standardized examination form will be used to determine the presence or absence of muscle weakness in a variety of muscle groups. The examination will be performed on arrival to the PACU and again 15 minutes after admission. Reported data is the total number of symptoms (0-16) at PACU admission
Time Frame: Early postoperative period, up to 24 hours
Measure: Median (Inter-Quartile Range); unit: symptoms
Arm/Group | Age 18-50 | Age 70-90
Number analyzed (Participants) | 150 | 149
symptoms | 2 [0 to 5] | 4 [1 to 8]

3. Secondary Outcome: Respiratory Events Potentially Related to Residual Neuromuscular Blockade
Description: Pulse oximetry will be used to continuously monitor arterial oxygen saturations (Sp02) during patient transport and in the PACU. Data reported are the number of patients developing hypoxemia (oxygen saturation < 94% on pulse oximetry) in the PACU
Time Frame: Early postoperative period, up to 24 hours
Measure: Number; unit: participants
Arm/Group | Age 18-50 | Age 70-90
Number analyzed (Participants) | 150 | 149
participants | 26 | 57

4. Secondary Outcome: PACU Length of Stay
Description: The time required to meet discharge criteria and achieve actual discharge will be noted.
Time Frame: Early postoperative period, up to 24 hours
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Age 18-50 | Age 70-90
Number analyzed (Participants) | 150 | 149
minutes | 73 [56 to 102] | 92 [67 to 125]

ADVERSE EVENTS:
Time Frame: Duration of hospitalization, which ranged from 1 to 10 days
Arm/Group | Age 18-50 | Age 70-90
Serious Adverse Events (participants affected / at risk) | 0/150 | 0/149
Other Adverse Events (participants affected / at risk) | 0/150 | 0/149

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes